CLINICAL TRIAL: NCT02265432
Title: iFit-Study: Using Mobile Technology to Promote Physical Activity
Brief Title: Using Mobile Technology to Promote Physical Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Falk Mueller-Riemenschneider (Other)
Responsible Party: Sponsor-Investigator, Dr Falk Mueller-Riemenschneider, Assistant Professor, National University of Singapore
Organization: National University of Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R -608-000-071-112
Record Dates: First submitted 2014-10-09; First posted 2014-10-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Physical Activity
Keywords: Physical activity; Sedentary behavior
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

ARMS (2):
- Mobile technology intervention (Experimental): 1. General physical activity educational materials
  2. Wearable activity tracking devices to enable the intervention participants to self-monitor their physical activity behavior and receive real-time feedback
  3. Access to an online map of Singapore providing location based information about leisure time physical activity opportunities
  4. Personalized text messages which include, educational information, tailored theory-based motivational messages, as well as compliance enhancing reminders
  Interventions: Behavioral: General physical activity educational materials; Device: Wearable activity tracking devices (fitbit); Other: online map; Other: Personalized text messages
- Control (Other): 1.General physical activity educational materials
  Interventions: Behavioral: General physical activity educational materials

INTERVENTIONS:
Behavioral: General physical activity educational materials
Device: Wearable activity tracking devices (fitbit)
  Arms: Mobile technology intervention
Other: online map
  Arms: Mobile technology intervention
Other: Personalized text messages
  Arms: Mobile technology intervention

SUMMARY:
The purpose of this study is to test an intervention which uses a personalized mobile-technology based approach that aims to promote physical activity and reduce sedentary behaviour in inactive working Singaporean adults.

DETAILED DESCRIPTION:
Considering the increasing burden in type 2 diabetes mellitus and other chronic diseases, the promotion of physical activity and reduction of sedentary behavior have an important role to improve population health.

Primarily, potential participants will be identified and recruited among participants from the Singapore Health Study (SHS) 2014 based on pre-specified selection criteria . SHS is a cross-sectional study of adults between 18 and 79 years which is conducted annually to monitor health, health behavior and health determinants among the Singapore general population.

All eligible participants will be randomized with a 1:1 ratio to intervention and control group.

Intervention group participants will receive a personalized mobile-technology based intervention to promote physical activity. It consists of four components:

1. General physical activity educational materials
2. Wearable activity tracking devices to enable the intervention participants to self-monitor their physical activity behavior and receive real-time feedback
3. Access to an online map of Singapore providing location based information about leisure time physical activity opportunities
4. Personalized text messages which include, educational information, tailored theory-based motivational messages, as well as compliance enhancing reminders

Control group participants will receive general physical activity educational materials, identical in content to that of the general educational materials of intervention group participants.

All participants will be assessed at baseline, 6 months and 12 months after the intervention by accelerometry and self-reported questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 25 to 65 years of age
* Physically inactive
* Working full-time for at least one more year after inclusion
* Signed written informed consent for the intervention study
* Willing to wear the activity tracker, fitbit all the time every day for 6 months

Exclusion Criteria:

* severe medical conditions prohibiting participation in physical activity
* pregnant women
* insufficient English language skills
* Participants who have already activity tracker device

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-04 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
average daily step counts | 6 months

SECONDARY OUTCOMES:
time spent in minutes per week on moderate- to vigorous- intensity physical activity measured by accelerometer | 6 months
time spent in sedentary activities per day | 6 months
level of physical activity(measured by accelerometer and self-report) determined in MET minutes per week | 6 months
time spent in vigorous-, moderate- and light- intensity activities will be determined. | 6 months

OTHER OUTCOMES:
proportion of participants being physical active according to current recommendations (at least 150 minutes of moderate intensity activity or an appropriate equivalent of vigorous activity) | 6 months
Recall, use and perceived usefulness of intervention and intervention components | 6 months
Knowledge, attitudes and perceived barriers to physical activity | 6 months
Quality of life | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Falk Mueller-Riemenschneider Falk <falk.mueller-riemenschneider, MSc, MD, Principal Investigator — Saw Swee Hock School of Public Health, National University of Singapore
Locations (1):
- National Univeristy of Singapore, Singapore, Singapore